CLINICAL TRIAL: NCT01167478
Title: Neurophysiological Reserve: Peripheral and Central Effects of Caffeine Manipulation
Brief Title: Neurophysiological Reserve With Caffeine Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Flavio de Oliveira Pires, Post-doctoral, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EEFE026; 2010/01317-0
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Caffeine; Placebo
Keywords: Exercise; Caffeine; Reserve
MeSH Terms: conditions — Motor Activity | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caffeine (Experimental)
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Caffeine — After ingestion of 6 mg.kg-1 of body mass of caffeine, subjects will perform the one exercise trial.
Dietary Supplement: Caffeine — 6 mg/kg of body mass of caffeine will be ingested by subjects before exercise.

SUMMARY:
The objective of this study is to verify if there is a neurophysiologic reserve when caffeine and placebo perceived as caffeine are manipulated in closed- and opened-loop exercises. Parameters of excitability level of skeletal muscle and Central Nervous System (CNS), and peripheral metabolism will be measured

DETAILED DESCRIPTION:
A neurophysiological reserve related to central mechanisms is supposed to be present, which should be observed when an increased central drive occurs. In theory, according to the central regulation model of effort, an increased performance could be due to the elevation on Central Nervous System excitability and activity, since exercise is not peripherally limited. Conversely, the absence of muscle performance improvement to the increased central drive promoted by caffeine would be an evidence for a peripherally localized neurophysiological limit and would indicate the absence of reserve. Therefore, if present, this reserve could be verified by using peripheral and central measures derived from electric-stimulation, evoked twitch and interpolated twitch techniques, associated to measures of EMG and peripheral metabolism, when caffeine is manipulated during closed- and opened-loop exercise.

In addition, there should also be possible to access the reserve without stimulant substance manipulation (placebo effect). By teleological argument derived from the central regulation model of effort, a neurophysiological reserve would be a natural mechanism to protect the cellular integrity. Therefore, it would be reasonable to hypothesize that, if present, a reserve would be observed by an increase in performance promoted by an elevation in central drive when placebo is perceived as caffeine. Unfortunately, however, no study utilized this experimental approach, including measures of central and peripheral activity during closed- and opened-loop exercise, to consistently respond the reserve question.

ELIGIBILITY:
Inclusion Criteria:

* trained cyclists
* trained in long distance races

Exclusion Criteria:

* Maximum oxygen uptake lower than 55 ml/kg/min

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Neurophysiological reserve evidenced by caffeine | Immediately after the administration (around 10 minutes)
  The time to cover a 4-km trial (closed-loop) or the time to exhaustion in an incremental intensity test (opened-loop) can show if the caffeine manipulation affects the performance. In addition, measures of CNS excitability such as EMG during the closed-loop exercise or at the exhaustion point in the opened-loop exercise, and measures such as the amplitude of H reflex, the rate of increase in H reflex/M wave relationship, can indicate if some central or peripheral alteration occurred during the exercises.
Neurophysiological reserve evidenced by caffeine | Immediately after the administration (around 10 minutes)
  The time to cover a 4-km trial (closed-loop) or the time to exhaustion in an incremental intensity test (opened-loop) can show if the placebo manipulation affects the performance. In addition, measures of CNS excitability such as EMG during the closed-loop exercise or at the exhaustion point in the opened-loop exercise, and measures such as the amplitude of H reflex, the rate of increase in H reflex/M wave relationship, can indicate if some central or peripheral alteration ocurred during the exercises.

SECONDARY OUTCOMES:
Neurophysiological reserve evidenced by placebo | Immediately after the administration (around 10 minutes)
  The placebo should also promote decrease in time of trial or increase in mean power output during a closed-loop exercise, elevation in time to exhaustion and maximal power output during an opened-loop exercise, and increase in maximal voluntary isometric contraction (MVIC) and time to contraction in a target force. Also, there should be a higher CNS excitability such as: 1) higher EMG during closed-loop exercise and higher EMG at the exhaustion point in an opened-loop exercise; 2) increased amplitude of H reflex; 3) elevation on the rate of increase in H reflex/M wave relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ugrinowitsch, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Lambert EV, St Clair Gibson A, Noakes TD. Complex systems model of fatigue: integrative homoeostatic control of peripheral physiological systems during exercise in humans. Br J Sports Med. 2005 Jan;39(1):52-62. doi: 10.1136/bjsm.2003.011247. PMID 15618343